CLINICAL TRIAL: NCT02920645
Title: Multicenter Validation of the AVICH Score
Acronym: AVICH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: AVICH-V1.1
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Intracerebral Hemorrhage; Arterio-venous Malformation
Keywords: ICH; AVM; intracerebral hemorrhage; arterio-venous malformation; AVICH
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AVM-related ICH patients: patients that suffered intracerebral hemorrhage (ICH) due to a ruptured artery-venous malformation (AVM)
  Interventions: Other: AVM-related ICH

INTERVENTIONS:
Other: AVM-related ICH

SUMMARY:
The primary objective of this multicenter study is to validate the AVICH score in terms of patient outcome prediction in AVM patients with associated ICH.

Secondary objectives are the impact of pretreatment of the AVICH score. Patients outcome is measured using the modified Rankin Scale (mRS) and are grouped in favorable (mRS score, 0-2) and unfavourable (mRS score, 3-6) outcome at last follow-up (LFU). The following parameters, which are part of the AVICH score, will be compared between the 2 groups: ICH score including age, Glasgow Coma Scale (GCS) score, haemorrhage volume, presence of intraventricular hemorrhage (IVH), and localization of the ICH. Spetzler-Martin grade including AVM size, eloquent location, and venous drainage, as well as the Lawton-Young grade, including age, presence of ruptured AVM, and the nidus structure. In addition pre-/postruptured treatment modalities, including embolization, radiotherapy, surgery or no treatment will be analysed. Outcome (mRS) at 3 months, at 1 year, and at LFU will be compared.

Multicentre validation study

Key inclusion criteria:

* All patients with ICH associated AVMs and a modified Rankin Scale <2 (so 0-1) before hemorrhage
* Pretreatment (embolization, radiosurgery, surgery) before ICH is not an exclusion criteria.

Key exclusion criteria:

* incomplete data set
* AVM Patients with only subarachnoid hemorrhage (SAH) or IVH and no ICH

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is the most common life threatening presentation of brain arteriovenous malformations (AVMs). Several AVM grading systems are available for presurgical risk assessment to help selecting patients for surgery. The most widely accepted and classic grading system is the Spetzler-Martin grading system; however, the recently introduced and externally validated supplemented Spetzler-Martin system seems to have an even better predictive accuracy. The pathophysiology of AVM-related ICH and spontaneous ICH is completely different. It is well known that clinical outcome in patients suffering spontaneous ICH is worse compared with patient outcome after AVM-related ICH. For spontaneous ICH, not related to AVM, several scoring systems exist to predict patient outcome. The most commonly used system is the ICH score. The available ICH scoring systems may not predict outcome in patients with hemorrhage caused by AVM rupture with the highest accuracy possible. Therefore, we examined a new scoring system called the AVM-related ICH score (AVICH score), which predicts patient outcome in the acute setting of AVM rupture. This scoring system is a special adaptation of the supplemented Spetzler-Martin grading system designed for patients presenting with hemorrhage, which includes additional clinical and radiographic information. Based on the area under the receiver operating characteristics curve (AUROC) analysis in this single center analysis, the AVICH score predicts outcome of patients with ruptured AVM and associated ICH better than the ICH score, the Spetzler-Martin, or the supplemented Spetzler-Martin grading system. An external validation is needed before the AVICH score is tested in a prospective multicenter cohort.

The primary objective of this multicenter study is to validate the AVICH score in terms of patient outcome prediction in AVM patients with associated ICH.

Secondary objectives are the impact of pretreatment of the AVICH score. Patients outcome is measured using the modified Rankin Scale (mRS) and are grouped in favorable (mRS score, 0-2) and unfavourable (mRS score, 3-6) outcome at last follow-up (LFU). The following parameters, which are part of the AVICH score, will be compared between the 2 groups: ICH score including age, Glasgow Coma Scale (GCS) score, haemorrhage volume, presence of intraventricular hemorrhage (IVH), and localization of the ICH. Spetzler-Martin grade including AVM size, eloquent location, and venous drainage, as well as the Lawton-Young grade, including age, presence of ruptured AVM, and the nidus structure. In addition pre-/postruptured treatment modalities, including embolization, radiotherapy, surgery or no treatment will be analysed. Outcome (mRS) at 3 months, at 1 year, and at LFU will be compared.

Key inclusion criteria:

* All patients with ICH associated AVMs and a modified Rankin Scale <2 (so 0-1) before hemorrhage
* Pretreatment (embolization, radiosurgery, surgery) before ICH is not an exclusion criteria.

Key exclusion criteria:

* incomplete data set
* AVM Patients with only SAH or IVH and no ICH

September, 1, 2016 - September, 30, 2016

* individual ethical approval each center (if needed)
* data collection (n = approximately 30/center)

November, 1, 2016 - November, 31, 2016

- data analysis (Zurich)

ELIGIBILITY:
Inclusion Criteria:

* All patients with ICH associated AVMs and a modified Rankin Scale <2 (so 0-1) before hemorrhage
* Pretreatment (embolization, radiosurgery, surgery) before ICH is not an exclusion criteria.

Exclusion Criteria:

* incomplete data set
* AVM Patients with only SAH or IVH and no ICH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that suffered from intracerebral hemorrhage (ICH) due to a ruptured artery-venous malformation (AVM)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
neurological long-term outcome (modified Ranking Scale, mRS) | up to 3 years at last follow-up

SECONDARY OUTCOMES:
neurological outcome (modified Ranking Scale, mRS) | 3 months after ICH
neurological outcome (modified Ranking Scale, mRS) | 1 year after ICH

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Karl Burkhardt, MD, Principal Investigator — Department of Neurosurgery, University Hospital Zurich, University of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neidert MC, Lawton MT, Mader M, Seifert B, Valavanis A, Regli L, Bozinov O, Burkhardt JK. The AVICH Score: A Novel Grading System to Predict Clinical Outcome in Arteriovenous Malformation-Related Intracerebral Hemorrhage. World Neurosurg. 2016 Aug;92:292-297. doi: 10.1016/j.wneu.2016.04.080. Epub 2016 May 2. PMID 27150647
- [Derived] Neidert MC, Lawton MT, Kim LJ, Nerva JD, Kurisu K, Ikawa F, Konczalla J, Dinc N, Seifert V, Habdank-Kolaczkowski J, Hatano T, Hayase M, Podlesek D, Schackert G, Wanet T, Glasker S, Griessenauer CJ, Ogilvy CS, Kneist A, Sure U, Seifert B, Regli L, Bozinov O, Burkhardt JK. International multicentre validation of the arteriovenous malformation-related intracerebral haemorrhage (AVICH) score. J Neurol Neurosurg Psychiatry. 2018 Nov;89(11):1163-1166. doi: 10.1136/jnnp-2017-316259. Epub 2017 Oct 6. PMID 28986471